CLINICAL TRIAL: NCT04361305
Title: Multicenter Study of the Efficacy and Safety of Dapoxetine Combined With Tadalafil in Men With Premature Ejaculation and Concomitant Erectile Dysfunction
Brief Title: Observational Study of Pharmacological Treatment for Premature Ejaculation Concurrent With Erectile Dysfunction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yan-Ping Huang (Other)
Responsible Party: Sponsor-Investigator, Yan-Ping Huang, Department of Urology and Andrology, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0412
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Premature Ejaculation; Erectile Dysfunction
MeSH Terms: conditions — Premature Ejaculation; Erectile Dysfunction | interventions — dapoxetine; Tadalafil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tadalafil combined with dapoxetine (Experimental)
  Interventions: Drug: Dapoxetine; Drug: Tadalafil
- tadalafil mono group (Active Comparator)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Dapoxetine — 30 mg tablets 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 8 weeks Tadalafil 5 mg tablets every day for 8 weeks
  Arms: tadalafil combined with dapoxetine
Drug: Tadalafil — 5 mg tablets every day for 8 weeks
  Arms: tadalafil mono group
Drug: Tadalafil — 5 mg tablets every day for 8 weeks
  Arms: tadalafil combined with dapoxetine

SUMMARY:
Premature ejaculation (PE) is a common disease in the andrology clinic. Currently, the effectiveness and outcome differences of drug treatment still need to be studied and demonstrated. Premature ejaculation concurrent with erectile dysfunction (ED) is common in outpatient clinics. The preferred treatment plan for these patients still needs to be further studied and explored, and the difference in the efficacy of different treatment regiments remain to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. PE concurrent with ED: the IELT is less than 3 minutes, the PEDT score is ≥11 points, and 5≤IIEF-5≤21 points.
2. 18-60 years old, outpatient or physical examination population, with regular sex partners and regular sex life;
3. Having the data below,and willing to participate in the trial（1）Demographic information: age, gender, nationality, birthplace, etc;(2) Physical examination data: height, weight, abdominal circumference, blood pressure, heart rate, etc ;(3) Medical history data: history of present illness, past medical history, family history, etc;(4) Scale evaluation: Premature Ejaculation Diagnostic Tool (PEDT), Premature Ejaculation Profile (PEP), International Erectile Function Score-5(IIEF-5), Erectile Hardness Grading Score (EHGS), Clinical Global Impression of Change (GICC);

Exclusion Criteria:

1. Age <18 years or> 60 years;
2. There is a history of acute and chronic diseases, major trauma and surgery, etc;
3. A long history of medication;
4. There is a history of unstable myocardial infarction and cerebral infarction;
5. A history of cardiogenic shock, severe heart failure, severe ventricular arrhythmia, etc;
6. There are serious diseases such as malignant tumors, chronic liver and kidney diseases, etc.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-03 (Estimated); Primary Completion 2021-01-11 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
The change of Premature Ejaculation Profile (PEP) at week 8 | Baseline, Week 8
  The PEP is a 4-question PRO that asks a respondent about his subjective sense of control over ejaculation, distress related to PE, interpersonal difficulty and satisfaction with sexual intercourse.
The change of International Index of Erectile Function -5(IIEF-5) at week 8 | Baseline, Week 8

SECONDARY OUTCOMES:
Incidence of adverse reactions | Baseline, Week 8
  To observe the safety of the two regiments in PE concurrent with ED patients
The change of Erection Hardness Score (EHS) | Baseline, Week 8
  Erection Hardness Score as a self-reporting measure that scored erection hardness on a 4 point scale. The aim was to help men, their partners and doctors diagnose erectile dysfunction.
Clinical Global Impression of Change (GICC) | Baseline, Week 8
  Clinical Global Impression is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.

IPD SHARING:
Plan to Share IPD: No